CLINICAL TRIAL: NCT02097342
Title: A Randomized Double-blind Study to Evaluate the Effect of Linagliptin on Pancreatic Beta Cell Function and Insulin Sensitivity in Patients With Type 2 Diabetes Mellitus on Metformin Monotherapy
Brief Title: Effect of Linagliptin on Insulin Sensitivity and Pancreatic Beta Cell Function in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Professor, Department of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Linagliptin
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Sensitivity/Resistance
Keywords: Type 2 Diabetes Mellitus; Insulin sensitivity- hyperinsulinemic euglycemic clamp; Pancreatic beta cell function; Linagliptin; Voglibose; Mixed meal test; GLP-1 response
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Linagliptin; voglibose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Linagliptin (Experimental): Tablet Linagliptin (5mg) per oral, once daily will be given to 10 patients for 6 months
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Tablet Placebo per oral, once daily will be given to 10 patients for 6 months
  Interventions: Drug: Placebo
- Voglibose (Active Comparator): Tablet Voglibose (0.2mg) per oral, thrice daily (with meals) will be given to 10 patients for 6 months
  Interventions: Drug: Voglibose

INTERVENTIONS:
Drug: Linagliptin — Tablet Linagliptin (5mg) per oral, once daily will be given to 10 patients for 6 months
  Other Names: Trajenta 5mg
  Arms: Linagliptin
Drug: Placebo — Tablet placebo per oral, once daily will be given to 10 patients for 6 months
  Arms: Placebo
Drug: Voglibose — Tablet Voglibose (0.2mg) per oral thrice daily(with meals) to 10 patients for 6 months
  Arms: Voglibose

SUMMARY:
This study is planned to evaluate if linagliptin can improve insulin sensitivity in patients with type 2 diabetes mellitus. In addition, the effect of linagliptin on pancreatic function will be studied.

DETAILED DESCRIPTION:
This is a prospective study of 30 patients with type 2 diabetes mellitus (T2DM) . Patients with T2DM in the age group 30-65 years and duration of diabetes less than five years will be screened. After exclusion, those who meet the inclusion criteria will be included in the study.

Once eligibility criteria are confirmed, patients will be educated about their disease and will be advised weight maintenance diabetic diet and exercise throughout the study period. Patients will be randomized to three groups - linagliptin (5mg OD) or voglibose (0.2mg TDS) or placebo OD. Metformin will be continued in all patients. To evaluate the effect of linagliptin on insulin sensitivity and beta cell function, independent of changes in HbA1c, the voglibose group is included. Each group will have 10 patients and will be followed up for 6 months. Both patients and physicians will be blinded to the treatment.

After having written informed consent, a detailed history and a thorough clinical examination will be done in all subjects including measurement of height, weight, body mass index and waist circumference. Hemoglobin, liver function tests, renal function tests, lipid profile, HbA1c, fasting plasma insulin , C-peptide, homeostasis model assessment-insulin resistance index(HOMA-1R) and homeostasis model assessment-beta cell function index (HOMA-β) will be done at baseline. A euglycemic hyperinsulinemic clamp study and a mixed meal test will be performed in all patients (on different days) at baseline and after 6 months of follow up. Biochemical parameters will be measured again 6 months after therapy. Fasting and post-prandial blood glucose will be done monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus (according to ADA guidelines)
* Age between 30-65 years
* Duration of diabetes less than five years
* BMI of between 20 and 40 kg/m2
* HbA1c level of < 7.5%
* On metformin monotherapy for at least 6 weeks

Exclusion Criteria:

* History of ketoacidosis
* Hepatic impairment (defined as plasma aminotransferase elevations of more than 3 times upper limit of normal)
* Renal failure (defined as Serum Creatinine more than 1.5 mg/dl)
* Coronary artery disease or heart failure
* Cerebrovascular disease or stroke
* Anemia (Hb< 10 g/dl)
* Those who requires insulin therapy HbA1c >7.5%
* Presence of macular edema
* Pregnant or lactating women
* Patients who have received dipeptidyl peptidase 4 (DPP-4) inhibitor therapy within last 3 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-11 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To study the effect of Linagliptin on insulin sensitivity by performing euglycemic hyperinsulinemic clamp in patients with type 2 diabetes mellitus. | 6 months
  Hyperinsulinemic euglycemic clamp of 2 hours duration will be done at baseline and after 6 months of treatment in all patients. Medications taken by the patient will be omitted on the day of test.After an overnight fast of 10 hours, intravenous catheter will be inserted, under sterile precautions, into the antecubital vein for infusion of insulin and dextrose solutions, while another catheter will be inserted in an anti-flow direction into the dorsal vein of the contralateral hand for arterialized blood sampling.
  An insulin infusate of 300 mU/ml will be administered at a constant rate, after an initial priming dose, while a 25 percent dextrose solution is administered at varying rates to maintain blood glucose at 90 mg/dl. Blood glucose will be analyzed by a bedside glucose analyzer every 5 minutes. M value, a measure of glucose utilisation will be calculated during the steady state (last 30 minutes of the test)

SECONDARY OUTCOMES:
To study the effects of Linagliptin on glycemic control and beta cell function in patients with type 2 diabetes mellitus 6 months | 6 months
  Fasting and 2 hour postprandial blood glucose will be at baseline and after 6 months of treatment. HbA1C will be done at baseline and after 3 and 6 months.
  HOMA-IR and HOMA-β will be done at baseline and after 6 months. Patients will also be subjected to a mixed meal test at baseline and at 6 months. Mixed meal test will be done 3-7 days after clamp study. After an overnight fast of 10 hours, patients will be given standardized mixed meal, 2.5 g/ kg. (Ensure, Abbott Nutrition, Abbott Laboratories) Medications normally taken by the subject in the morning will be administered 20 min prior to the start of the test meal. Samples for glucose, insulin, C-peptide and glucagon-like peptide-1 (GLP-1) will be taken at 0,30,60,90,120,150 and 180 minutes following the ingestion of meal. Total area under curves for glucose, insulin, C-peptide and GLP-1 from pre meal to 180 min will be calculated using the trapezoidal rule.

OTHER OUTCOMES:
To study the effect of voglibose on glucagon like peptide1 (GLP1) secretion and insulin resistance in patients with type 2 diabetes mellitus 6 months | 6 months
  Patients will be subjected to mixed meal test and a hyperinsulinemic euglycemic clamp study at baseline and after 6 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education & Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Parthan G, Bhansali S, Kurpad AV, Walia R, Bhat K, Bhansali A. Effect of Linagliptin and Voglibose on metabolic profile in patients with Type 2 Diabetes: a randomized, double-blind, placebo-controlled trial. BMC Pharmacol Toxicol. 2018 Jul 3;19(1):38. doi: 10.1186/s40360-018-0228-z. PMID 29970184